CLINICAL TRIAL: NCT04121299
Title: Mechanism of Masked Hypertension - Intervention
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mohammed Siddiqui, MD, Postdoctoral Fellow, Vascular Biology and Hypertension Program, Division of Cardiovascular Disease, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300004152
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Masked Hypertension
Keywords: Masked Hypertension; Sympathetic Activity; Sympatholytic Therapy
MeSH Terms: conditions — Masked Hypertension | interventions — Carvedilol; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carvedilol 40mg Extended Release Once Daily (Experimental): participants will be randomized to carvedilol 40 mg extended release once daily for the 1st or 2nd 4 week treatment period
  Interventions: Drug: Carvedilol
- Amlodipine 10mg Once Daily (Active Comparator): participants will be randomized to amlodipine 10 mg once daily for the 1st or 2nd 4 week treatment period
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Carvedilol — Carvedilol 40mg Extended Release Once Daily
  Arms: Carvedilol 40mg Extended Release Once Daily
Drug: Amlodipine — Amlodipine 10mg Once Daily
  Arms: Amlodipine 10mg Once Daily

SUMMARY:
To test the hypothesis that sympatholytic antihypertensive antihypertensive therapy (αβ-blocker - carvedilol) will reduce out-of-clinic ambulatory BP to a greater extent by blocking sympathetic activity than non-sympatholytic antihypertensive medication (dihydropyridine calcium channel blocker - amlodipine) in individuals with masked hypertension.

DETAILED DESCRIPTION:
A. Participants. Study participants with masked hypertension (MH) with controlled clinic BP (< 130/80 mmHg) and uncontrolled out-of-clinic awake ambulatory BP (ABP ≥ 130/80 mmHg) untreated with antihypertensive medications will be recruited.

B. Study design. This is a double-blinded, randomized, 2-period, 2-treatment crossover clinical trial comparing sympatholytic antihypertensive agent (αβ-blocker - carvedilol 40mg extended release once daily) with non-sympatholytic control agent (dihydropyridine calcium channel blocker - amlodipine 10mg once daily) in individuals with MH. All study participants will undergo out-of-clinic 24hr ABP with actigraphy monitoring for 24-hr, awake and asleep ABP; sympathetic activity assessment by BP and HR variability, 24-hour urinary catecholamines and metanephrines at baseline and after intervention. In order to avoid selection bias, patients will be randomized to their initial therapy. Patients and study personnel will be blinded to the treatment group in order to minimize information bias. An investigator without direct study involvement will be assigned the task of ensuring correct dispensing of the study medication, which will be prepared as matching capsules by the UAB Pharmacy - Investigational Drug Service. After 4 weeks of initial treatment, both treatment groups will undergo a 1-month washout where no study medication is given in order to prevent a carryover effect. The study medication will be taken in the morning between 6 and 9 am except for study visit days. A crossover design is chosen to minimize differences between study groups, as participants will act as their own controls. Electrolytes, kidney function and ECG will be monitored at each visit. Medication adherence will be determined at visit 2 (week 4) and visit 4 (week 12) by measuring 24-hr urinary specimens for medications and their metabolites by LC-MS/MS and by pill count and medication log.

C. Outcomes. The primary outcome is the difference in percent change in out-of-clinic mean 24-hr ABP, awake ABP and asleep ABP with carvedilol compared to amlodipine. Secondary outcomes include change in out-of-clinic sympathetic activity by BP and HR variability; and 24-hour urinary catecholamines and metanephrines.

D. Preliminary / anticipated results. We anticipate a greater reduction in out-of-clinic 24-hr, awake and asleep ABP due to blocking of sympathetic activity with carvedilol when compared to amlodipine use in individuals with MH. A statistically significant effect estimate will support our hypothesis that higher sympathetic activity contributes to MH, which can be managed by use of sympatholytic agents like carvedilol.

ELIGIBILITY:
Study participants with masked hypertension i.e. controlled clinic blood pressure (BP) and uncontrolled out-of-clinic awake ambulatory BP will be enrolled.

A. Inclusion criteria.

* Adults (18-75 years of age)
* Controlled clinic BP (< 130/80 mmHg) untreated with antihypertensive medications
* Uncontrolled awake ambulatory BP (≥ 130/80 mmHg) untreated with antihypertensive medications

B. Exclusion criteria.

* Hypertensive (Clinic BP ≥ 130/80 mmHg)
* Hypotensive (Clinic BP < 90/70 mmHg)
* Bradycardic (Heart rate < 60 beats/minute)
* Heart block
* Use of an antihypertensive medication within the last 3 months
* Use of an steroid containing medications within the last 3 months
* Body mass index ≥ 30 Kg/m2
* Chronic kidney disease (Estimated GFR < 60 mL/min/1.73m2)
* Primary aldosteronism
* Renal artery stenosis
* Pheochromocytoma
* Diabetes mellitus
* Pregnant women
* Breast feeding women
* Dementia and/or cognitive impairment prohibiting consent
* History of stroke within the past 6 months
* History of unstable angina within the past 6 months
* History of myocardial infarction within the past 6 months
* Allergy or intolerance to β-blockers
* Allergy or intolerance to calcium channel blockers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Out of clinic 24 hour ambulatory blood pressure | 4 weeks
  Difference in percent change in out-of-clinic mean 24-hr ambulatory BP in mmHg with carvedilol compared to amlodipine.
Out of clinic awake blood pressure | 4 weeks
  Difference in percent change in out-of-clinic mean awake ambulatory BP in mmHg with carvedilol compared to amlodipine.
Out of clinic asleep blood pressure | 4 weeks
  Difference in percent change in out-of-clinic mean asleep ambulatory BP in mmHg with carvedilol compared to amlodipine.

SECONDARY OUTCOMES:
Out of clinic blood pressure variability | 4 weeks
  Change in out-of-clinic sympathetic activity by BP variability in mmHg with carvedilol compared to amlodipine.
Out of clinic heart rate variability | 4 weeks
  Change in out-of-clinic sympathetic activity by HR variability in beats/minute with carvedilol compared to amlodipine.
Out of clinic 24-hour urinary catecholamines | 4 weeks
  Change in out-of-clinic sympathetic activity by 24-hour urinary catecholamines levels with carvedilol compared to amlodipine.
Out of clinic 24-hour urinary metanephrines | 4 weeks
  Change in out-of-clinic sympathetic activity by 24-hour urinary metanephrines levels with carvedilol compared to amlodipine.

CONTACTS AND LOCATIONS:
Locations (1):
- Hypertension Research Clinic at UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Will adhere to the NIH Data Sharing and Implementation policy:
  https://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm
  Data Sharing: Unpublished research data will be presented at scientific meetings. These regularly include American Heart Association Council on Hypertension Scientific Sessions and Southern Society of Clinical Investigators-southern regional meeting. Moreover, unpublished data, including methodologies and datasets will be uploaded to RedCap with access granted to mentor, co-mentors and members of mentoring committee. All data acquired will be shared and made publicly available through publication in the peer-reviewed literature.
Time Frame: Research data will be shared with non-participating investigators once the data are accepted for publication.
Access Criteria: All accepted manuscripts will be submitted electronically to PubMed Central (PMC) via the NIH Manuscript Submission (NIHMS) system according to journal policy and NIH agreements. Through the Freedom of Information Act, the data in the publications and the raw data documents will be made available upon written request.